CLINICAL TRIAL: NCT04059484
Title: An Open Label Randomized Phase 2 Trial of Amcenestrant (SAR439859), Versus Endocrine Monotherapy as Per Physician's Choice in Patients With Estrogen Receptor-positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer With Prior Exposure to Hormonal Therapies
Brief Title: Phase 2 Study of Amcenestrant (SAR439859) Versus Physician's Choice in Locally Advanced or Metastatic ER-positive Breast Cancer
Acronym: AMEERA-3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT16105; U1111-1217-2774 (Registry Identifier: ICTRP); 2018-004593-98 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — Fulvestrant; Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amcenestrant (Experimental): Daily amcenestrant dose administered orally under fed or fast condition
  Interventions: Drug: Amcenestrant
- Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator (Active Comparator): Control treatment of the choice of the physician depending on each participant's medical condition and in accordance with the approved label may include 1 of the following treatments used as monotherapy.
  Fulvestrant
  Aromatase inhibitors (anastrozole, letrozole, exemestane)
  Selective estrogen receptor modulator (Tamoxifen)
  Interventions: Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Tamoxifen

INTERVENTIONS:
Drug: Amcenestrant — Pharmaceutical form: Capsule
  Route of administration: Oral
  Arms: Amcenestrant
Drug: Fulvestrant — Pharmaceutical form: Solution for injection
  Route of administration: Intramuscular
  Other Names: Faslodex®
  Arms: Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator
Drug: Anastrozole — Pharmaceutical form:Tablets or capsules
  Route of administration: Oral
  Other Names: Arimidex®/Anastrozole Generics
  Arms: Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator
Drug: Letrozole — Pharmaceutical form: Tablets or capsules
  Route of administration: Oral
  Other Names: Femara®/Letrozole Generics
  Arms: Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator
Drug: Exemestane — Pharmaceutical form: Tablets or capsules
  Route of administration: Oral
  Other Names: Aromasin®/Exemestane Generics
  Arms: Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator
Drug: Tamoxifen — Pharmaceutical form: Tablets or capsules
  Route of administration: Oral
  Other Names: Nolvadex®/Tamoxifen Generics
  Arms: Fulvestrant/Aromatase inhibitors/Estrogen receptor modulator

SUMMARY:
Primary Objective:

To determine whether amcenestrant per overall survival (os) improves progression free survival (PFS) when compared with an endocrine monotherapy of the choice of the physician, in participants with metastatic or locally advanced breast cancer

Secondary Objectives:

* To compare the overall survival in the 2 treatment arms
* To assess the objective response rate in the 2 treatment arms
* To evaluate the disease control rate in the 2 treatment arms
* To evaluate the clinical benefit rate in the 2 treatment arms
* To evaluate the duration of response in the 2 treatment arms
* To evaluate the PFS according to the estrogen receptor 1 gene (ESR1) mutation status in the 2 treatment arms
* To evaluate the pharmacokinetics of amcenestrant as single agent
* To evaluate health-related quality of life in the 2 treatment arms
* To compare the overall safety profile in the 2 treatment arms

DETAILED DESCRIPTION:
The duration of the study for an individual participant will include a period to assess eligibility (screening period) of up to 4 weeks (28 days), a treatment period of at least 1 cycle (28 days of study treatment), and an end of treatment (EOT) visit at least 30 days (or until the participant receive another anticancer therapy, whichever is earlier) following the last administration of study treatment. Study treatment may continue until precluded by unacceptable toxicity, disease progression, death or upon participant's request to stop treatment, or Investigator decision, whichever occurs first.

An extension of recruitment for Chinese participants is planned in this study: After completion of randomization in the global part of the study, randomization will continue in China until approximately 90 Chinese participants are randomized.

ELIGIBILITY:
Inclusion criteria :

* 18 years or older.
* Histological or cytological diagnosis of adenocarcinoma of the breast.
* Locally advanced not amenable to radiation therapy or surgery in a curative intent, and/or metastatic disease.
* Estrogen receptor(ER) positive status.
* Human epidermal growth factor receptor 2 negative status.
* Participants must have received no more than 1 prior chemotherapeutic or 1 targeted therapy regimen for advanced/metastatic disease.
* In the main study, a prior treatment with a Cyclin-dependent kinase 4 and 6(CDK 4/6) inhibitor is mandatory if this treatment is approved and can be reimbursed for this participant. The percentage of participants without previous CDK 4/6 inhibitor will be capped to 20%. In the Chinese extension cohort, previous treatment with a CDK 4/6 inhibitor will not be mandatory, and there will be no limitation to the number of participants naïve to CDK4/6 inhibitor.
* Participants must present a secondary endocrine resistance to endocrine therapy defined as: progression while on endocrine therapy after at least 6 months of treatment for advanced breast cancer, or relapse while on adjuvant endocrine therapy but after the first 2 years, or with a relapse within 12 months after completing adjuvant endocrine therapy.
* Male or Female.

Exclusion criteria:

* Eastern Cooperative Oncology Group performance status =>2.
* Medical history or ongoing gastrointestinal disorders potentially affecting the absorption of amcenestrant. Participants unable to swallow normally and to take capsules.
* Participant with any other cancer. Adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or any other cancer from which the participant has been disease free for greater than 3 years are allowed.
* Severe uncontrolled systemic disease at screening .
* Participants with known brain metastases that are untreated, symptomatic or require therapy to control symptoms.
* Prior treatment with mammalian target of rapamycin inhibitors or any other selective estrogen receptor degrader(SERD) compound, except fulvestrant if stopped for at least 3 months before randomization.
* Treatment with drugs that have the potential to inhibit Uridine'5 Diphospho-Glucuronosyl Transferase(UGT) less than 2 weeks before randomization.
* Treatment with strong Cytochrome P450 (CYP)3A inducers within 2 weeks before randomization.
* Ongoing treatment with drugs that are sensitive substrate of organic anion transporting polypeptide 1B1/B3(OATP1B1/B3) (asunaprevir, atorvastatin, bosentan, danoprevir, fexofenadine, glyburide, nateglinide, pitavastatin, pravastatin, replaglinide, rosuvastatin, and simvastatin acid).
* Treatment with anticancer agents (including investigational drugs) less than 3 weeks before randomization.
* Inadequate hematological, coagulation, renal and liver functions.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2025-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (109):
- United States (14):
  - Alabama Oncology Site Number : 8400008, Birmingham, Alabama
  - Comprehensive Blood and Cancer Center Site Number : 8400018, Bakersfield, California
  - UCLA Hematology Oncology Parkside Site Number : 8400024, Santa Monica, California
  - The University of Kansas Clinical Research Center Site Number : 8400027, Fairway, Kansas
  - Hematology Oncology Clinic Site Number : 8400020, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute Site Number : 8400015, Boston, Massachusetts
  - Saint Luke's Hospital Site Number : 8400032, Kansas City, Missouri
  - Dartmouth Hitchcock Med Center Site Number : 8400013, Lebanon, New Hampshire
  - Hackensack University Medical Center Site Number : 8400025, Hackensack, New Jersey
  - Gabrail Cancer Center Site Number : 8400006, Canton, Ohio
  - The Center For Cancer And Blood Disorders Site Number : 8400022, Fort Worth, Texas
  - University Of Vermont Site Number : 8400026, Burlington, Vermont
  - Northwest Medical Specialties Site Number : 8400038, Tacoma, Washington
  - University of Wisconsin Site Number : 8400016, Madison, Wisconsin
- Argentina (7):
  - Investigational Site Number : 0320008, CABA, Buenos Aires
  - Investigational Site Number : 0320007, Capital Federal, Buenos Aires
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320004, La Rioja
  - Investigational Site Number : 0320002, Salta
- Australia (3):
  - Investigational Site Number : 0360003, South Brisbane, Queensland
  - Investigational Site Number : 0360002, Woolloongabba, Queensland
  - Investigational Site Number : 0360001, Nedlands, Western Australia
- Belgium (3):
  - Investigational Site Number : 0560002, Charleroi
  - Investigational Site Number : 0560001, Leuven
  - Investigational Site Number : 0560003, Namur
- Brazil (5):
  - Hospital Araujo Jorge Site Number : 0760005, Goiânia, Goiás
  - Hospital de Clinicas de Porto Alegre - HCPA Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Hospital de Base Sao Jose do Rio Preto Site Number : 0760003, São José do Rio Preto, São Paulo
  - Nucleo de Pesquisa Clinica e Ensino da Rede Sao Camilo Site Number : 0760006, São Paulo, São Paulo
- Canada (3):
  - Investigational Site Number : 1240004, Calgary, Alberta
  - Investigational Site Number : 1240003, London, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
- China (18):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560015, Changchun
  - Investigational Site Number : 1560014, Changsha
  - Investigational Site Number : 1560025, Chengdu
  - Investigational Site Number : 1560024, Chongqing
  - Investigational Site Number : 1560023, Hangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560005, Harbin
  - Investigational Site Number : 1560010, Hefei
  - Investigational Site Number : 1560018, Hefei
  - Investigational Site Number : 1560026, Jinan
  - Investigational Site Number : 1560003, Kunming
  - Investigational Site Number : 1560008, Linyi
  - Investigational Site Number : 1560011, Nanjing
  - Investigational Site Number : 1560013, Tianjin
  - Investigational Site Number : 1560021, Ürümqi
  - Investigational Site Number : 1560016, Wuhan
  - Investigational Site Number : 1560031, Xuzhou
- Czechia (3):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030003, Nový Jičín
  - Investigational Site Number : 2030004, Prague
- France (5):
  - Investigational Site Number : 2500008, Angers
  - Investigational Site Number : 2500006, Créteil
  - Investigational Site Number : 2500007, Marseille
  - Investigational Site Number : 2500005, Paris
  - Investigational Site Number : 2500001, Villejuif
- Greece (3):
  - Investigational Site Number : 3000001, Heraklion
  - Investigational Site Number : 3000002, Larissa
  - Investigational Site Number : 3000004, Thessaloniki
- Israel (4):
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760003, Tel Aviv
  - Investigational Site Number : 3760004, Tel Litwinsky
- Italy (3):
  - Investigational Site Number : 3800001, Candiolo, Torino
  - Investigational Site Number : 3800002, Milan
  - Investigational Site Number : 3800003, Prato
- Japan (8):
  - Investigational Site Number : 3920002, Nagoya, Aichi-ken
  - Investigational Site Number : 3920001, Kashiwa-shi, Chiba
  - Investigational Site Number : 3920009, Ota-shi, Gunma
  - Investigational Site Number : 3920006, Yokohama, Kanagawa
  - Investigational Site Number : 3920003, Osaka, Osaka
  - Investigational Site Number : 3920005, Kitaadachi-gun, Saitama
  - Investigational Site Number : 3920004, Chuo-ku, Tokyo
  - Investigational Site Number : 3920008, Koto-ku, Tokyo
- Latvia (2):
  - Investigational Site Number : 4280002, Riga
  - Investigational Site Number : 4280001, Riga
- Mexico (3):
  - Investigational Site Number : 4840002, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, México
  - Investigational Site Number : 4840006, Veracruz
- Poland (2):
  - Investigational Site Number : 6160003, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
- Torre Hospital Auxilo Mutuo Site Number : 8400028, Ponce de Leon 735 Hato Rey, Puerto Rico, Puerto Rico
- Russia (3):
  - Investigational Site Number : 6430003, Moscow
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430002, Saint Petersburg
- South Korea (4):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240008, Málaga
- Taiwan (5):
  - Investigational Site Number : 1580002, Taichung
  - Investigational Site Number : 1580003, Tainan
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580005, Taipei
  - Investigational Site Number : 1580004, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920004, Ankara
  - Investigational Site Number : 7920002, Edirne
  - Investigational Site Number : 7920003, Istanbul
- Ukraine (3):
  - Investigational Site Number : 8040001, Kryvyi Rih
  - Investigational Site Number : 8040004, Odesa
  - Investigational Site Number : 8040005, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Tolaney SM, Chan A, Petrakova K, Delaloge S, Campone M, Iwata H, Peddi PF, Kaufman PA, De Kermadec E, Liu Q, Cohen P, Paux G, Wang L, Ternes N, Boitier E, Im SA. AMEERA-3: Randomized Phase II Study of Amcenestrant (Oral Selective Estrogen Receptor Degrader) Versus Standard Endocrine Monotherapy in Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer. J Clin Oncol. 2023 Aug 20;41(24):4014-4024. doi: 10.1200/JCO.22.02746. Epub 2023 Jun 22. PMID 37348019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 88 active centers in 22 countries. A total of 366 participants were screened between 22 October 2019 and 15 April 2021 in the global cohort, of which 76 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 290 participants were randomized in the study. Randomization was stratified according to presence of visceral metastasis (defined by at least 1 liver or lung metastasis; yes or no), prior treatment with a cyclin-dependent kinase 4/6 (CDK4/6) inhibitors (yes/no), and Eastern Cooperative Oncology Group (ECOG) status (0 or 1). Assignment to the arms was done in a 1:1 ratio using interactive response technology (IRT). Results reported based on primary completion date of 15 February 2022.
Groups:
- Physician Choice Endocrine Monotherapy (PCEM): Participants received potential control treatment of the choice of the physician depending on each participant's medical condition and in accordance with the approved label. Control treatment included one of the following treatments to be selected before randomization and used as monotherapy: 1) Fulvestrant 500 milligrams (mg), given as two 5-milliliters (mL) intramuscular (IM) injections on Cycle 1 Days 1 and 15, and at Day 1 of each 28-day treatment cycle thereafter; or 2) Aromatase inhibitors (anastrozole 1 mg or letrozole 2.5 mg or exemestane 25 mg) orally (PO), once a day (QD); or 3) Tamoxifen 20 mg/day PO, QD or twice a day (maximum exposure: 116 weeks).
- Amcenestrant: Participants received 4 capsules of 100 mg, amcenestrant PO, QD from Day 1 to Day 28 in each 28-day treatment cycle until precluded by unacceptable toxicity or disease progression or participant's request to stop treatment or Investigator decision, whichever occurred first (maximum exposure: 116 weeks).
Period: Overall Study
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Started | 147 | 143
Completed | 0 | 0
Not Completed | 147 | 143
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Progressive disease | 112 | 112
Not completed — Other | 8 | 3
Not completed — Ongoing | 20 | 20

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) population which included all enrolled participants (i.e., who sign the informed consent form [ICF]) and for whom there is a confirmation of successful allocation of a randomization number by IRT.
Groups:
- Physician Choice Endocrine Monotherapy (PCEM): Participants received potential control treatment of the choice of the physician depending on each participant's medical condition and in accordance with the approved label. Control treatment included one of the following treatments to be selected before randomization and used as monotherapy: 1) Fulvestrant 500 mg, given as two 5-mL IM injections on Cycle 1 Days 1 and 15, and at Day 1 of each 28-day treatment cycle thereafter; or 2) Aromatase inhibitors (anastrozole 1 mg or letrozole 2.5 mg or exemestane 25 mg), PO, QD; or 3) Tamoxifen 20 mg/day PO, QD or twice a day (maximum exposure: 116 weeks).
- Total: Total of all reporting groups
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant | Total
Number analyzed (Participants) | 147 | 143 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.5) | 58.2 (11.8) | 58.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 143 | 289
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 32 | 66
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 0 | 0 | 0
  White | 102 | 102 | 204
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in months interval from the date of randomization to the date of first documented tumor progression as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) assessed by independent central review (ICR) or death (due to any cause), whichever comes first. Progressive Disease (PD) as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the date of first documented tumor progression or death due to any cause or data cut-off date whichever comes first (maximum duration: 116 weeks)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Physician Choice Endocrine Monotherapy (PCEM): Participants received potential control treatment of the choice of the physician depending on each participant's medical condition and in accordance with the approved label. Control treatment included one of the following treatments to be selected before randomization and used as monotherapy: 1) Fulvestrant 500 mg, given as two 5-mL IM injections on Cycle 1 Days 1 and 15, and at Day 1 of each 28-day treatment cycle thereafter; or 2) Aromatase inhibitors (anastrozole 1 mg or letrozole 2.5 mg or exemestane 25 mg) PO, QD; or 3) Tamoxifen 20 mg/day PO, QD or twice a day (maximum exposure: 116 weeks).
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
months | 3.7 [2.0 to 4.9] | 3.6 [2.0 to 3.9]
Statistical Analysis 1: Comparison: Physician Choice Endocrine Monotherapy (PCEM) vs Amcenestrant; A hierarchical testing procedure was used to ensure a strong control of the overall Type I error. Testing was then performed sequentially in order the outcome measures was reported and continued when previous outcome measure was statistically significant at one-sided 2.5% for the primary and the first secondary outcome; Test type: Superiority; p = 0.6437, Stratified Log-Rank test — One-sided p-value based on Stratified log-rank test. Threshold for statistical significance at 0.025 level; Stratified on presence of visceral metastasis, prior treatment with CDK4/6 inhibitors and ECOG according to IRT; Hazard Ratio (HR) = 1.051, 95% CI 2-sided [0.789 to 1.4] — Amcenestrant versus PCEM

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from the date of randomization to the date of documented death (due to any cause). In the absence of observation of death, survival time was censored to last date the participant is known to be alive or at the cut-off date, whichever comes first. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the death due to any cause or data cut-off date whichever comes first (maximum duration: 116 weeks)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
months | NA [18.9 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to the smaller number of participants with events. | NA [21.5 to NA] — Median and upper limit of 95% CI was not estimable due to the smaller number of participants with events.

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response is defined as percentage of participants having a partial response (PR) or complete response (CR) according to the RECIST version 1.1 assessed by ICR. As per RECIST 1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to the date of first documented tumor progression, death due to any cause or data cut-off date whichever comes first (maximum duration: 116 weeks)
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
percentage of participants | 8.8 [4.8 to 14.6] | 11.9 [7.1 to 18.4]

4. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control is defined as percentage of participants having a confirmed CR, PR, or stable disease (SD) or Non-CR/Non-PD as BOR determined by ICR as per RECIST 1.1 from the date of randomization to the date of end of treatment. As per RECIST 1.1, CR: disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters. Non-CR/Non-PD: persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 3
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
percentage of participants | 53.7 [45.3 to 62.0] | 54.5 [46.0 to 62.9]

5. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical Benefit is defined as percentage of participants having a confirmed CR, PR, SD, or Non-CR/Non-PD for at least 24 weeks determined by ICR as per RECIST 1.1 from the date of randomization to the date of end of treatment. As per RECIST 1.1, CR: disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters. Non-CR/Non-PD: persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 3
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
percentage of participants | 29.3 [22.0 to 37.3] | 27.3 [20.2 to 35.3]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as time (in months) from first documented evidence of CR or PR until progressive disease (PD) determined by ICR as per RECIST 1.1 or death from any cause, whichever occurs first. For participants with ongoing response at the time of the analysis, DOR was censored at the date of the last valid disease assessment not showing documented progression performed before the initiation of a new anticancer treatment (if any). As per RECIST 1.1, CR: disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions.
Time Frame: From the date of first response to the date of first documented tumor progression, death due to any cause or data cut-off date whichever comes first (maximum duration: 116 weeks)
Population: Analysis was performed on a subset of participants who had objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 13 | 17
months | NA [3.9 to NA] — Median and upper limit of 95%CI was not estimable due to the small number of progression events or death. | 15.1 [5.6 to NA] — Upper limit of 95%CI was not estimable due to small number of progression events or death.

7. Secondary Outcome: Progression Free Survival (PFS) According to Estrogen Receptor 1 Gene (ESR1) Mutation Status
Description: PFS defined as the time (in months) interval from the date of randomization to the date of first documented tumor progression as per RECIST 1.1 assessed by ICR or death (due to any cause), whichever comes first. Progression as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. The mutation status (wild type, mutant) of twelve specific mutations of the ESR1 gene was determined by multiplex droplet digital polymerase chain reaction (ddPCR), including their mutant frequency and concentration. Here, PFS is reported based on the ESR1 mutation status of participants: wild type and mutants. ESR1 was the gene encoding estrogen receptor alpha. ESR1 mutant type breast cancer was a disease where the ESR1 gene had a mutation (i.e., a type of error). ESR1 wild type breast cancer was a disease where the ESR1 gene was normal without a mutation. Analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Analysis was performed on the ITT population. Here, "overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" = participants with available data for each specified category.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Amcenestrant: Participants received 4 capsules of 100 mg, PO of amcenestrant QD from Day 1 to Day 28 in each 28-day treatment cycle until precluded by unacceptable toxicity or disease progression or participant's request to stop treatment or Investigator decision, whichever occurred first (maximum exposure: 116 weeks)
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 140 | 140
months
  Mutated: number analyzed (Participants) | 55 | 65
  Mutated | 2.0 [1.9 to 4.3] | 3.7 [1.9 to 7.2]
  Wild type: number analyzed (Participants) | 85 | 75
  Wild type | 3.9 [3.6 to 9.2] | 3.5 [2.0 to 3.7]

8. Secondary Outcome: Pharmacokinetics: Plasma Concentrations of Amcenestrant
Description: Amcenestrant plasma concentrations at specified time points are reported.
Time Frame: Cycle 1 Day 1: 1.5 hours(h), 4h post-dose, Day 15: pre-dose, Cycle 2 Day 1: pre-dose, 1.5h, 4h, 8h post-dose, Cycle 3 Day 1: pre-dose, Cycle 4 Day 1: pre-dose, Cycle 6 Day 1: pre-dose
Population: Analysis was performed on Pharmacokinetic-evaluable population: all participant who were assigned to study intervention, took at least 1 dose of study intervention, had at least 1 available plasma concentration post treatment with adequate documentation of date and time of dosing and date and time of sampling. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for PCEM group arm.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Amcenestrant
Number analyzed (Participants) | 140
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: 1.5h: number analyzed (Participants) | 130
  Cycle 1 Day 1: 1.5h | 3185.7 (3145.2)
  Cycle 1 Day 1: 4h: number analyzed (Participants) | 128
  Cycle 1 Day 1: 4h | 4753.1 (3463.7)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 87
  Cycle 1 Day 15: Pre-dose | 516.4 (377.2)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 98
  Cycle 2 Day 1: Pre-dose | 479.1 (320.3)
  Cycle 2 Day 1: 1.5h: number analyzed (Participants) | 121
  Cycle 2 Day 1: 1.5h | 2719.6 (2374.0)
  Cycle 2 Day 1: 4h: number analyzed (Participants) | 115
  Cycle 2 Day 1: 4h | 3801.8 (2370.8)
  Cycle 2 Day 1: 8h: number analyzed (Participants) | 98
  Cycle 2 Day 1: 8h | 2303.8 (1411.4)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 42
  Cycle 3 Day 1: Pre-dose | 593.6 (815.1)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 44
  Cycle 4 Day 1: Pre-dose | 661.5 (860.5)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 28
  Cycle 6 Day 1: Pre-dose | 531.5 (468.5)

9. Secondary Outcome: Within-Participant Steady State Ctrough of Amcenestrant
Description: Within-participant Steady state Ctrough was defined as the median value of the Ctrough across study using plasma concentration of predose samples at Cycle 1 Day 15 and Day 1 of Cycle 2, 3, 4 and 6 for each individual participant. Average (mean) of all calculated Ctrough values for all participants across study (Cycle 1 Day 15 and Day 1 of Cycle 2, 3, 4 and 6 ) was derived and reported in this outcome measure.
Time Frame: Predose on Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4 Day 1; Cycle 6 Day 1
Population: Analysis was performed on Pharmacokinetic-evaluable population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for PCEM group arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amcenestrant
Number analyzed (Participants) | 123
ng/mL | 491.35 (316.51)

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) Domain Scores
Description: EORTC-QLQ-C30: cancer-specific instrument with 30 questions for evaluation of new chemotherapy & assessment of participant reported outcome. These include 5 functional scales, 9 symptom scales, & Global Health Status/quality of life scale (GHS/QoL). All 14 items/domains were scored on scale of 1 (not at all) to 4 (very much) and GHS/QoL, scored on scale of 1 (very poor) to 7 (excellent). All scales are transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional & GHS/QoL = higher level of functioning, & higher score for symptoms scales = higher symptom burden. Least Square (LS) mean and Standard Error (SE) are derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 30]) was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 30 [i.e.,116 weeks])
Population: Analysis was performed on safety population evaluable which includes all participants randomly assigned to study intervention, who took at least 1 dose of study intervention, completed the baseline and at least 1 post baseline on-treatment assessment. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Physician Choice Endocrine Monotherapy (PCEM): Participants received potential control treatment of the choice of the physician depending on each participant's medical condition and in accordance with the approved label. Control treatment included one of the following treatments to be before randomization and used as monotherapy: 1) Fulvestrant 500 mg, given as two 5-mL IM injections on Cycle 1 Days 1 and 15, and at Day 1 of each 28-day treatment cycle thereafter; or 2) Aromatase inhibitors (anastrozole 1 mg or letrozole 2.5 mg or exemestane 25 mg) PO, QD; or 3) Tamoxifen 20 mg/day PO, QD or twice a day (maximum exposure: 116 weeks).
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
score on a scale
  GHS/QoL: number analyzed (Participants) | 130 | 125
  GHS/QoL | 1.8 (1.6) | 2.5 (1.6)
  Physical functioning: number analyzed (Participants) | 131 | 126
  Physical functioning | -1.2 (1.3) | -3.1 (1.3)
  Role functioning: number analyzed (Participants) | 131 | 126
  Role functioning | -2.4 (1.9) | -3.0 (1.8)
  Emotional functioning: number analyzed (Participants) | 131 | 126
  Emotional functioning | -2.2 (1.7) | 3.0 (1.6)
  Cognitive functioning: number analyzed (Participants) | 131 | 126
  Cognitive functioning | -0.9 (1.6) | -0.8 (1.5)
  Social functioning: number analyzed (Participants) | 130 | 126
  Social functioning | -2.5 (1.7) | -0.8 (1.7)
  Fatigue: number analyzed (Participants) | 131 | 126
  Fatigue | 1.1 (1.9) | 2.8 (1.9)
  Nausea and vomiting: number analyzed (Participants) | 131 | 126
  Nausea and vomiting | 1.7 (1.3) | 1.3 (1.3)
  Pain: number analyzed (Participants) | 131 | 126
  Pain | 1.1 (1.9) | 2.1 (1.9)
  Dyspnoea: number analyzed (Participants) | 131 | 125
  Dyspnoea | 1.0 (1.6) | 0.8 (1.6)
  Insomnia: number analyzed (Participants) | 131 | 126
  Insomnia | -1.1 (2.3) | -2.3 (2.2)
  Appetite loss: number analyzed (Participants) | 130 | 126
  Appetite loss | 2.4 (2.3) | 1.2 (2.3)
  Constipation: number analyzed (Participants) | 131 | 126
  Constipation | -2.3 (2.0) | 3.0 (2.0)
  Diarrhoea: number analyzed (Participants) | 130 | 126
  Diarrhoea | 0.3 (1.3) | 3.9 (1.3)
  Financial difficulties: number analyzed (Participants) | 131 | 126
  Financial difficulties | 1.7 (1.8) | -2.0 (1.8)

11. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions (5D), 5 Levels (5L) (EQ-5D-5L) Score: Visual Analog Scale (VAS) Score
Description: EQ-5D-5L is a standardized measure of health status, provides a simple, generic measure of health for clinical and economic appraisal, and consists of 2 sections: the EQ-5D-5L health state utility index (descriptive system) and the EQ-5D-5L VAS. The Visual Analogue Scale is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. LS mean and SE are derived from MMRM model with change from baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from Baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 30]) was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 30 [i.e.,116 weeks])
Population: Analysis was performed on Safety population evaluable. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 125 | 125
score on a scale | 0.9 (1.4) | 0.2 (1.4)

12. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions (5D), 5 Levels (5L) (EQ-5D-5L) Score: Health Utility Index Value
Description: EQ-5D-5L: consists of 2 sections: EQ-5D-5L health state utility index (descriptive system) & VAS. The EQ-5D descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, & extreme problems. Response options are measured with 5-point Likert scale (for 5L version). The EQ-5D-5L responses are converted into single index utility score between 0 to 1, where higher score indicates better health state & lower score indicate worse health state. LS mean and SE are derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from baseline values overall treatment (i.e., each cycle [Cycle 1 up to Cycle 30]) was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 30 [i.e.,116 weeks])
Population: Analysis was performed on Safety population evaluable. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 124 | 129
score on a scale | -0.0 (0.0) | -0.0 (0.0)

13. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Breast Cancer Specific Module (EORTC-QLQ-BR23) Domain Scores
Description: QLQ-BR23: disease-specific Health-related QOL assesses impact of breast cancer & side effects of treatment. EORTC-QLQ-BR23 contains 23 items: multi-item scales & single-item measures. 4 functional scales (body image, sexual functioning, sexual enjoyment, future perspective) & 4 scales related to symptoms of disease or treatment (arm symptoms, breast symptoms, systemic therapy side effects, & upset by hair loss). All items scored 1 (not at all) to 4 (very much). Scores of all scales transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional scales = better outcome; higher score for symptoms scales = higher symptom burden. LS mean and SE are derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 30]) was reported.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 30 [i.e.,116 weeks])
Population: Analysis was performed on Safety population evaluable. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant
Number analyzed (Participants) | 147 | 143
score on a scale
  Body image: number analyzed (Participants) | 132 | 130
  Body image | 1.8 (1.7) | 2.2 (1.6)
  Sexual functioning: number analyzed (Participants) | 127 | 127
  Sexual functioning | -2.4 (1.3) | -2.6 (1.2)
  Sexual enjoyment: number analyzed (Participants) | 33 | 20
  Sexual enjoyment | -1.1 (3.0) | 0.4 (4.1)
  Future perspective: number analyzed (Participants) | 132 | 130
  Future perspective | 10.6 (2.7) | 12.0 (2.6)
  Systemic therapy side effects: number analyzed (Participants) | 133 | 130
  Systemic therapy side effects | 0.2 (1.0) | 0.7 (1.0)
  Breast symptoms: number analyzed (Participants) | 129 | 128
  Breast symptoms | -0.4 (1.3) | -0.8 (1.2)
  Arm symptoms: number analyzed (Participants) | 130 | 128
  Arm symptoms | 1.8 (1.7) | 2.0 (1.7)
  Upset by hair loss: number analyzed (Participants) | 37 | 47
  Upset by hair loss | -9.7 (3.9) | -10.6 (3.7)

ADVERSE EVENTS:
Time Frame: AE data was collected from Baseline up to 30 days after the last treatment administration (up to a maximum of 116 weeks), deaths were collected from Baseline up to the cut-off date (15 February 2022)
Description: Reported adverse events (AEs) are treatment-emergent AEs that developed, worsened, or became serious during the treatment period (time from the first dose of study treatments up to 30 days after last dose of study treatments). Serious and Other AEs were collected for safety population only. All-Cause Mortality data collected during the study was assessed for all randomized participants. Disease progression related death were not reported as AE.
Groups:
- Amcenestrant 400 mg: Participants received 4 capsules of 100 mg, amcenestrant PO, QD from Day 1 to Day 28 in each 28-day treatment cycle until precluded by unacceptable toxicity or disease progression or participant's request to stop treatment or Investigator decision, whichever occurred first (maximum exposure: 116 weeks).
Arm/Group | Physician Choice Endocrine Monotherapy (PCEM) | Amcenestrant 400 mg
All-Cause Mortality (participants affected / at risk) | 2/147 | 5/143
Serious Adverse Events (participants affected / at risk) | 15/147 | 23/143
Other Adverse Events (participants affected / at risk) | 76/147 | 84/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Choice Endocrine Monotherapy (PCEM) (N=147) | Amcenestrant 400 mg (N=143)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 0 (0)
Peritonitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Contrast Media Allergy (Immune system disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 2 (2) | 4 (4)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Respiratory Distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Choice Endocrine Monotherapy (PCEM) (N=147) | Amcenestrant 400 mg (N=143)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 10 (11)
Headache (Nervous system disorders) | 14 (14) | 18 (19)
Hot Flush (Vascular disorders) | 13 (13) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (8)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 14 (17)
Nausea (Gastrointestinal disorders) | 13 (14) | 28 (34)
Vomiting (Gastrointestinal disorders) | 5 (5) | 27 (43)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 20 (24)
Back Pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 18 (20)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (9)
Asthenia (General disorders) | 8 (8) | 11 (16)
Fatigue (General disorders) | 17 (18) | 16 (18)
Injection Site Pain (General disorders) | 10 (20) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04059484/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04059484/SAP_001.pdf